CLINICAL TRIAL: NCT05293210
Title: Early Treatment Strategy With High-dose Dexamethasone Versus Standard Dose in Patients With SARS-CoV-2 Pneumonia (COVID-19). PREDEXACOV Study
Brief Title: Early Treatment Strategy With High-dose Dexamethasone in Patients With SARS-CoV-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDEXACOV
Record Dates: First submitted 2021-04-26; First posted 2022-03-24 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Dexamethasone
Keywords: dexamethasone; covid19
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: The study consists of 2 phases:
  * Hospitalization phase: Day 1 of IC signature to day of hospital discharge. In case of not having completed 10 days of hospitalization since inclusion, patients will have to complete the 10 days of treatment on an outpatient basis. This medication will be provided by the Hospital Pharmacy. In case of discharge, the information will be obtained from the patients in person or by telephone contact, according to their needs, with the patient himself or his caregivers and/or cohabitants.
  * Follow-up phase: outpatient visits at 30, 60 and 90 days. The information is obtained from the patients, from the medical records or by telephone contact with the patient himself or his caregivers and/or cohabitants according to availability and need of the patient.
Masking Description: Patients who meet all inclusion criteria and none of the exclusion criteria will be randomized to receive a daily dose of dexamethasone 20 mg intravenous for 3 days, followed by a daily dose of oral or intravenous dexamethasone 6 mg for 7 more days versus the center's standard treatment which includes the use of oral or intravenous dexamethasone 6 mg for 10 days with escalation to a daily dose of oral or intravenous dexamethasone 20 mg for 3 days if clinical criteria of respiratory distress develop despite treatment with dexamethasone 6 mg daily.
  Randomization will be performed in a centralized manner. Randomization will be done directly in the database itself by including the patient in the CRD-e (Redcap). When the investigator registers a patient in the CRD-e, the system will directly assign him/her to which group he/she has been randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): A daily dose of dexamethasone 20 mg intravenous for 3 days, followed by a daily dose of dexamethasone 6 mg intravenous or oral for 7 days.
  Interventions: Drug: Dexamethasone
- Standard treatment regimen (Active Comparator): Dexamethasone 6 mg orally or intravenously for 10 days (with the possibility of escalation to doses of 20 mg daily of oral or intravenous dexamethasone for 3 days if clinical criteria of respiratory distress develop despite treatment with doses of dexamethasone 6 mg daily).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — A daily dose of dexamethasone 20 mg intravenous for 3 days, followed by a daily dose of dexamethasone 6 mg intravenous or oral for 7 days.
  Dexamethasone 6 mg orally or intravenously for 10 days (with the possibility of escalation to doses of 20 mg daily of oral or intravenous dexamethasone for 3 days if clinical criteria of respiratory distress develop despite treatment with doses of dexamethasone 6 mg daily).

SUMMARY:
Early identification and treatment of this inflammatory cascade using existing therapeutic strategies with proven safety profiles could change the course and prognosis of COVID-19 infection, reducing mortality rates. Glucocorticoids may modulate inflammation-mediated lung injury and thereby reduce progression to respiratory failure and death

DETAILED DESCRIPTION:
The use of corticosteroids in COVID 19 in hospitalized patients with moderate symptoms has not been adequately studied in randomized clinical trials, the studies and clinical trials having focused on critical or severe patients. The few studies available to date have yielded evidence of low certainty.

Our trial postulates that early intervention and treatment with high-dose corticosteroids (20 mg dexamethasone for 3 days) in patients admitted with pneumonia with respiratory failure and moderate elevation of acute phase reactants and proinflammatory cytokines, or with risk factors that condition worse prognosis on admission, and who have not yet developed data on respiratory distress, the development of the cytokine storm could be avoided or minimized, reducing lung tissue damage and progression to severe respiratory failure and, therefore, reducing the need for invasive and noninvasive respiratory therapies, reducing hospital stay and, possibly, reducing associated mortality.

Dexamethasone is a potent synthetic glucocorticoid with actions resembling those of steroid hormones. It acts as an anti-inflammatory and immunosuppressant. It is a widely known glucocorticoid, studied and used in the treatment of autoimmune diseases, in oncology patients under chemotherapy to counteract certain side effects of their antitumor treatment, to augment the antiemetic effects of 5-HT3 receptor antagonists, in patients with brain neoplasms (primary or metastatic) to reduce edema, in spinal cord compressions, in certain hematological malignancies, in the treatment of arthropathies, to counteract allergic shock and septic shock, among many other indications for use. It is also used for the diagnosis of diseases related to hypothalamic-pituitary-adrenal axis dysfunction.

Recently, following the DEXA-COVID, CoDEX and RECOVERY clinical trials, dexamethasone has been widely used in patients with severe or critical SARS-CoV-2 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with SARS-CoV-2 (COVID19) pneumonia confirmed by antigenic test or PCR Age ≥ 18 yrs.
* pcr ≥ 66 mg/L and ≤150 mg/L at inclusion or Pandemic score at admission > 200 with pcr 9.7-149 mg/L at inclusion.
* WHO scale level 4, with need for oxygen therapy in NG ≥ 1 lpm to maintain saturation ≥ 94%.
* Onset of symptoms ≤ 10 days before the date of inclusion.
* After having received verbal and written information about the study, the patient must submit the signed and dated Informed Consent before performing any activity related to the study.

Exclusion Criteria:

* Patients with respiratory distress criteria at the time of randomization, understood as need for OCNAF/VMNI/VMI (levels 5 and 6 of the WHO scale) or O2 saturation ≤ 92% and/or FR ≥ 30 despite oxygen in NG at 4 liters.
* Patients with allergy or contraindication to the use of systemic corticosteroids.
* Patients with severe asthma or chronic pulmonary pathology with home oxygen requirements and active treatment with corticosteroids.
* Patients on chronic corticosteroid treatment.
* Use of corticosteroids daily in the 15 days prior to hospital admission.
* Indication of corticosteroid use due to other clinical conditions of the patient (e.g., septic shock).
* Pregnant or actively breastfeeding women
* Patients with suspected or confirmed bacterial, fungal, or viral infection other than SARS-CoV-2 itself at the time of randomization
* Patients with confirmed past or latent tuberculosis infection prior to inclusion.
* Patients with known HIV infection with CD4 below 500 cells/mm3 or on active treatment with protease inhibitors or boosters such as cobicistat or ritonavir.
* Patients with active oncologic processes in the last year or in active treatment with chemotherapy.
* Patients with life expectancy < 3 months at inclusion due to clinical conditions other than SARS-CoV-2 pneumonia.
* Patients with expected death in the following 48-72 hours.
* Patients included in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate if there is a decrease in the proportion of patients who develop respiratory distress | Week 12
  * To evaluate whether there is a decrease in the proportion of patients who develop respiratory distress with the need for NIV/MIV/OCNAF (measured group and individually by respiratory therapies).
  * To evaluate the impact of this strategy on the number of days of hospitalization.

SECONDARY OUTCOMES:
Evaluate if there is a decrease in the number of therapy days | W12
  * To evaluate whether there is a decrease in the number of NIV/MIV/OCNAF therapy days.
  * To evaluate whether there is a decrease in all-cause mortality at 30, 60 and 90 days.
  * Safety: short- and long-term adverse events related to the following

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carranza, MD, Principal Investigator — Infanta Leonor University Hospital